CLINICAL TRIAL: NCT02988908
Title: Memory and Mental Health in Aging: Psychopharmacological Augmentation of Memory Training in Older Adults
Brief Title: Memory and Mental Health in Aging
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jerome A Yesavage,, Principle Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SU-06302009-2820; R01MH035182 (NIH); eprotocol #7530 (Other: Stanford University)
Record Dates: First submitted 2010-05-11; First posted 2016-12-09 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2016-12

CONDITIONS: Memory
MeSH Terms: interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug: Donepezil (Experimental): Participants received Donepezil as 5mg pills per day for 6 weeks, then 10 mg per day for the remainder of the 52-week trial.
  Participants also received 2 weeks of memory training at weeks 13-14
  Interventions: Drug: Donepezil
- Placebo (Control) (Placebo Comparator): Participants received placebo as 5mg pills per day for 6 weeks, then 10 mg per day for the remainder of the 52-week trial.
  Participants also received 2 weeks of memory training at weeks 13-14
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Donepezil — Participants received donepezil as 5mg pills per day for 6 weeks, then 10 mg per day for the remainder of the 52-week trial.
  Participants also received 2 weeks of memory training at weeks 13-14
  Other Names: Aricept
  Arms: Drug: Donepezil
Drug: Placebos — Participants received placebo as 5mg pills per day for 6 weeks, then 10 mg per day for the remainder of the 52-week trial.
  Participants also received 2 weeks of memory training at weeks 13-14
  Other Names: Control
  Arms: Placebo (Control)

SUMMARY:
A comparison of memory training with and without donepezil.

DETAILED DESCRIPTION:
Study 1:

Investigators evaluated the short-term and longer-term efficacy and effectiveness of a pharmacologic augmentation strategy for a nonpharmacologic treatment to improve memory performance in nondemented older adults. Investigators used a randomized controlled trial with parallel groups design that compares two Treatments: DONEPEZIL + COGNITIVE TRAINING versus PLACEBO + COGNITIVE TRAINING.

Study 2:

The second study looked more closely at dosage. Investigators hoped to determine the best dosage of the drug donepezil for enhancing the effects of the memory training program.

ELIGIBILITY:
Inclusion Criteria:

Study 1 only:

1. Global Clinical Dementia Rating (CDR) 0.0 or 0.5, at least 1 Box score = 0.5 and none > 0.5;
2. Laboratory normal B12, RPR, and Thyroid Function Tests or without any clinically significant abnormalities that would be expected to interfere with the study, plus general clinical chemistry and complete blood count.
3. ECG without clinically significant abnormalities that would be expected to interfere with the study

Study 1 and Study 2:

1. Mini-Mental Exam score between 24 and 30 (inclusive);
2. General cognition and functional performance sufficiently preserved such that a diagnosis of Alzheimer's Disease cannot be made by the site physician at the time of the screening visit;
3. Permitted medications stable for at least 1 month prior to screening. In particular: a) Subjects may take stable doses of antidepressants lacking significant anticholinergic side effects (if they are not currently depressed and do not have a history of major depression within the past 2 years). b) Estrogen replacement therapy is permissible. c) Ginkgo biloba is permissible, but discouraged.
4. Hamilton Depression Score less than or equal to 12 on the 17-item scale.
5. Visual and auditory acuity adequate to allow neuropsychological testing.
6. General health good with no additional diseases expected to interfere with the study.
7. Women two years post-menopausal or surgically sterile.

Exclusion Criteria:

1. Any significant neurologic disease such as Possible and Probable AD, Parkinson's disease, multi-infarct dementia, Huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma followed by persistent neurologic defaults or known structural brain abnormalities.
2. Major depression or another major psychiatric disorder as described in DSM IV within the past 2 years. History of schizophrenia (DSM IV criteria). Psychotic features, agitation or behavioral problems within the last 3 months which could lead to difficulty complying with the protocol.
3. History of alcohol or substance abuse or dependence within the past 2 years (DSM IV criteria).
4. Any significant systemic illness or unstable medical condition which could lead to difficulty complying with the protocol including:

   1. History of systemic cancer within the last 5 years (non-metastatic skin cancers are acceptable).
   2. History of myocardial infarction within the past year or unstable or severe cardiovascular disease including angina or CHF with symptoms at rest.
   3. Clinically significant obstructive pulmonary disease or asthma.
   4. Clinically significant and unstable gastrointestinal disorder such as ulcer disease or a history of active or occult gastrointestinal bleeding within two years.
   5. Insulin-requiring diabetes or uncontrolled diabetes mellitus.
   6. Uncontrolled hypertension (systolic BP greater than 170 or diastolic greater than 100).
   7. History of clinically significant liver disease, coagulopathy, or vitamin K deficiency within the past 2 years.
5. Use of centrally active beta-blockers, narcotics, methyldopa and clonidine within 4 weeks prior to screening. b) Use of anti-Parkinsonian medications (e.g. Sinemet, amantadine, bromocriptine, pergolide and selegiline) within 2 months prior to screening. c) Use of neuroleptics or narcotic analgesics within 4 weeks prior to screening. d) Use of long-acting benzodiazepines or barbiturates within 4 weeks prior to screening. e) Use of short-acting anxiolytics or sedative hypnotics more frequently than 2 times per week within 4 weeks prior to screening (note: sedative agents should not be used within 72 hours of screening). f) Initiation or change in dose of an antidepressant lacking significant cholinergic side effects within the 4 weeks prior to screening (use of stable doses of antidepressants for at least 4 weeks prior to screening is acceptable). g) Use of systemic corticosteroids within 3 months prior to screening. h) Medications with significant cholinergic or anticholinergic side effects (e.g. pyridostigmine, tricyclic antidepressants, meclizine, and oxybutynin) within 4 weeks prior to screening. i) Use of anti-convulsants (e.g. Phenytoin, Phenobarbital, Carbamazepine) within 2 months prior to screening. j) Use of warfarin (Coumadin) within 4 weeks prior to screening.
6. Any prior use of any FDA approved medications for the treatment of Alzheimer's Disease (e.g. tacrine, donepezil, or other newly approved medications).
7. Use of any investigational drugs within 30 days or 5 half-lives, whichever is longer, prior to screening.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2000-04; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Change in recall of Word List over time | measured at baseline, Week 13 (before training), Week 14 (at end of training), and Week 52
  Each participant was given a list of 16 words. Participants had 4 minutes to memorize the words in order. Short-term recall was tested after 5 minutes exposure to a distractor task and delayed recall was tested after 30 minutes. At recall participants were asked to recall as many words as they could remember in the order the words were presented.
Change in recall of Name-Face pairs over time | measured at baseline, Week 13 (before training), Week 14 (at end of training), and Week 52
  Each participant was shown 12 name-face pairs for 1 minute. Recall was tested immediately after presentation of all 12 name-face pairs (faces were shown for 1 minute and participant was asked to supply the name).

SECONDARY OUTCOMES:
Change in Symbol Digit score over time | measured at baseline, Week 13, and Week 52
  Symbol Digit modalities test (Smith 1991)
Change in Digit Span score over time | measured at baseline, Week 13, and Week 52
  Digit Span from the Wechsler, 1987
Change in Medical Outcomes Study Functioning and Well-being Profile over time | measured at baseline, Week 13, and Week 52
  Measuring Functioning and Well-Being is a comprehensive account of a broad range of self-reported functioning and well-being measures developed for the Medical Outcomes Study (Stewart AL, 1992)
Change in Everyday Problems Test score over time | measured at baseline, Week 13 (before training), and Week 52
  Measure of Functional Capacity (Willis SL, Mariske M, 1993)

CONTACTS AND LOCATIONS:
Overall Officials: Jerome A Yesavage, Principal Investigator — Stanford University
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No